CLINICAL TRIAL: NCT05753280
Title: Effect of Serum Vitamin D Level and Vitamin D Receptor on the Efficacy of Pegylated Interferon in Patients With Chronic Hepatitis B With Low Level HBsAg Treated by Nucleos(t)Ide Analogues
Brief Title: Effect of Serum Vitamin D Level on the Efficacy of Peg-interferon Treatment in CHB
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Third Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Zhiliang Gao, Academic leader of the infectious diseases department, Third Affiliated Hospital, Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: G58
Record Dates: First submitted 2023-02-22; First posted 2023-03-03 (Actual); Last update posted 2023-03-03 (Actual); Status verified 2023-02

CONDITIONS: Chronic Hepatitis b
Keywords: hepatitis B; Vitamin D; Interferon
MeSH Terms: conditions — Hepatitis B, Chronic; Hepatitis B | interventions — Vitamin D

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- treatment group (Experimental): pegylated interferon 180ug/week and oral vitamin D3 800IU/day for no longer than 48 weeks
  Interventions: Drug: Vitamin D
- control group (No Intervention): pegylated interferon 180ug/week for no longer than 48 weeks

INTERVENTIONS:
Drug: Vitamin D — Patients take 800 mg vitamin D capsules daily during the whole treatment period
  Arms: treatment group

SUMMARY:
In recent years, vitamin D (VD) has received much attention in the fields of host immune regulation, inflammation, fibrosis, cell proliferation and differentiation and tumor. VD works by binding to the vitamin D receptor (VDR). VDR is mainly distributed in giant cells, dendritic cells, T cells and lymphocytes. Four SNPs of VDRS have been most studied: TaqI (rs731236), FokI (rs10735810), ApaI (rs7975232), and BsmI (rs1544410). At present, more and more patients have been treated with oral nucleotide/nucleoside analogues (NAs) with direct antiviral drugs in China, and a large part of them show low expression of HBsAg. Clinical cure can be pursued for these patients, that is, HBsAg turns negative. A number of studies have been carried out at home and abroad.

In this study, We will recruit CHB patients with low HBsAg levels. They all will receive pegylated interferon treatment and were randomly assigned to a vitamin D treatment or a control group. A final assessment will be made to determine whether vitamin D levels would affect the clearance rate of HBsAg.

ELIGIBILITY:
Inclusion Criteria:

1.According with the diagnosis of chronic hepatitis B in the guideline of China in 2015 2.18-60 years old 3.More than 1 year history of nucleot(s)ide analogues therapy with HBsAg ≤1500 IU/ml, negative HBeAg and HBV DNA<100 IU/ml 4.No contraindications of interferon

Exclusion Criteria:

1. Allergy to interferon
2. Alanine transaminase >10 times of upper limit of normal(ULN) or total bilirubin >2 times of ULN
3. existing or previous decompensated liver cirrhosis
4. White blood cells or Platelet below the lower limit of normal
5. existing severe organ injury
6. combined with autoimmune diseases, psychiatric diseases, diabetes or thyroidism
7. confirmed or suspected malignant tumors
8. before or after transplantation
9. using immunosuppressor
10. pregnant or having a planned parenthood in 2 years
11. alcohol or drug addicted
12. infected by HIV
13. any conditions that is unsuitable to interferon therapy according to the doctors' judgement

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
hepatitis B surface antigen | up to 48 weeks
  hepatitis B surface antigen should be tested by the reagents from Roche or Abbott, which is expressed by using IU/ml.

SECONDARY OUTCOMES:
hepatitis B surface antibody | every 12 weeks for up to 48 weeks
  hepatitis B surface antigen should be tested by the reagents from Roche or Abbott, which is expressed by using IU/ml

CONTACTS AND LOCATIONS:
Overall Officials: Zhiliang Gao, Doctor, Study Chair — Third Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- Department of Infectious Diseases, The Third Affliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No